CLINICAL TRIAL: NCT06985251
Title: CommitFit App to Facilitate Health Behavior Change in Clinic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Amy Braddock, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2092610
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Overweight Adolescents
Keywords: mHealth; obesity; adolescent; parent; caregiver; financial incentives; behavior modification; user engagement
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CommitFit$ (Experimental): Adolescents in CommitFit$ were paid $0.05 for each point they earned when using app
  Interventions: Other: gamified mHealth app with financial incentives
- CommitFit (Experimental): Caregivers and Adolescents using CommitFit app without additional financial incentives
  Interventions: Other: gamified mHealth lifestyle app
- Control (Active Comparator): Attention, wait-list controls were emailed monthly healthy lifestyle handouts and were allowed to download CommitFit after 4 month study period ended.
  Interventions: Other: Attention Control

INTERVENTIONS:
Other: gamified mHealth lifestyle app — The CommitFit mHealth app uses gamification techniques to motivate adolescents and caregivers to set and achieve health behavior goals (eat more fruits or vegetables, increase water intake, decrease sugary beverage intake, increase physical activity, or increase overnight sleep). Users are ranked on leaderboard based on their points and can team up with caregivers on a team leaderboard.
  Arms: CommitFit
Other: Attention Control — Standard of care healthy lifestyle handouts were emailed monthly to control families.
  Arms: Control
Other: gamified mHealth app with financial incentives — The CommitFit mHealth app uses gamification techniques to motivate adolescents and caregivers to set and achieve health behavior goals (eat more fruits or vegetables, increase water intake, decrease sugary beverage intake, increase physical activity, or increase overnight sleep). Users are ranked on leaderboard based on their points and can team up with caregivers on a team leaderboard. CommitFit$ adolescents received an extra $0.05 for each point they earned in the app.
  Arms: CommitFit$

SUMMARY:
We conducted a 3-month RCT with 30 adolescents (aged 13-15 years) and their caregivers to evaluate the effectiveness of the novel mHealth app "CommitFit", which uses gamification to motivate users to log and achieve health behavior goals. The RCT had three arms: (1) CommitFit only users, (2) CommitFit$, adolescents were paid $0.05 for each point they earned, and (3) Control. Software analytics, surveys, BMI, and blood pressure were evaluated at baseline, 3 months, and 4 months.

DETAILED DESCRIPTION:
We will recruit 30 adolescents and 30 caregivers to beta test CommitFit. The study will be limited to one participating adolescent and one of their caregivers. There will be three groups in the study: 1) Control 2) CommitFit and 3) CommitFit$.

All participants will be required to complete a screening survey at the beginning of the study. The eligible participants will be contacted via email/ phone and will give their consent after taking the screening survey, and then they will take the baseline demographic survey for their adolescents and themselves.

After the participants in the CommitFit and CommitFit$ groups download the app, they will be shown how to pick a health behavior (fruits/vegetables, water, decreased sugary beverages, physical activity, sleep) and then set a goal and a time period to work on their goal. They will receive a daily reminder to log their health behaviors. At the end of their goal period, they will be rewarded with points for logging behaviors and successfully achieving their goals. Points will be used to rank the participant on the leaderboard using the username that they registered with. Users can also use points to unlock gear for their avatar in the gear store. Control group participants will receive email handouts with healthy lifestyle tips which they could use if they choose to. They will not use the CommitFit app. All participants will be compensated through eGift cards.

Software analytics will be utilized to evaluate how the app was used (frequency of goals set and behaviors logged), duration of use, etc., to evaluate app features and gamification techniques. We will evaluate changes in health behaviors using online surveys, and measure health metrics (height and weight which will be used to calculate Body Mass Index (BMI), and blood pressure) in the clinic.

We will have the adolescents take 7 surveys-GAD7, PedQL, Reasons why I think about being healthy, Behavior economics survey, Gamification Survey, CommitFit App Survey, and Commercialization Survey (CommitFit and CommitFit$ only for use surveys). Similarly, we will have the caregivers take 4 surveys Gamification Survey, CommitFit App Survey, Behavior economics survey, and Commercialization Survey for caregiver subject. In the control group, adolescents will only take 4 surveys- GAD7, PedQL, Reasons why I think about being healthy, and Behavior economics survey. Caregivers in the control group will take only the Behavioral Economic survey. All participants will take the surveys at the beginning of the study, after end of 3rd month, and at the end of the 4th month (follow-up visit). Weight, height and blood pressure from all adolescents and their caregivers will also be collected at the clinical site. All participants completed the 5-10 minute paper exit survey and interview at their final 4-month clinic visit.

ELIGIBILITY:
Inclusion Criteria: speak English fluently, read at the 6th grade level or higher, and be proficient with smart phone app use to participate. Caregivers much bet at least 18 years or older. No baseline weight criteria.

-

Exclusion Criteria: severe mental health disorders (other than mild or controlled anxiety and/or depression), intellectual disabilities, or eating disorders via a screening survey

-

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
BMI percentile | Baseline to 4 months
  Change in BMI percentile for adolescents

SECONDARY OUTCOMES:
BMI | Baseline to 4 months
  Change in BMI in adult caregivers
%goal achieved | Baseline to 4 months
  Number of times the user achieved their self-selected health behavior goal divided by the number of possible times they could have achieved health behavior goal. Users can achieve up to 2 goals per day, every day.

OTHER OUTCOMES:
%logged | Baseline to 4 months
  How of then user logged a health behavior goal in CommitFit app divided by how often they could have logged. Users can log up to 2 goals per day, each day.
blood pressure | Baseline to 4 months
  blood pressure in adolescents and caregivers
GAD7 | Baseline to 4 months
  anxiety in adolescents
PedQL | Baseline to 4 months
  Pediatric Quality of Life in adolescents
Reasons why I think about being healthy | Baseline to 4 months
  Health behavior motivation survey in adolescent
CommitFit surveys | Baseline to 4 months
  Surveys developed by the research team to evaluate CommitFit app including behavior economics, gamification, app use survey, and commercialization in adolescents and caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- South Providence Medical Park, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include survey data, analytic data generated from the mHealth CommitFit app software, anthropometrics (height, weight, blood pressure, waist circumference), and survey data. To protect the identities of participants, all data will be deidentified before final storage and sharing.
Supporting Information: Study Protocol
Time Frame: Start date will be upon publication of primary outcomes, anticipated to be 1/1/2026. There will be no end date as deidentified data will be available permanently through the data repository at the University of Missouri (MOspace Institutional Repository)
Access Criteria: All data will be shared within IRB and HIPAA-approved parameters. The PI will monitor and restrict access of identified data to IRB-approved staff. Deidentified data submitted to MOspace will be publicly accessible
URL: https://mospace.umsystem.edu/xmlui/

REFERENCES:
- [Background] Braddock A, Ghosh P, Montgomery E, Lim C, Ghosh J, Henry N, Popescu M, Kimchi K, Guo C, Bosworth KT, Koopman RJ. Effectiveness of an mHealth App That Uses Financial Incentives and Gamification to Promote Health Behavior Change in Adolescents and Caregivers: Protocol for a Clinic-Based Randomized Controlled Trial. JMIR Res Protoc. 2024 Sep 10;13:e63505. doi: 10.2196/63505. PMID 39255473
- [Derived] Henry N, Montgomery E, Ghosh P, Bosworth KT, Lim C, Ghosh J, Popescu M, Kimchi K, Guo C, Smith J, Braddock A. Caregiver inclusion influence on adolescent acceptance and engagement of an mHealth app, a randomized controlled trial. Mhealth. 2025 Oct 29;11:57. doi: 10.21037/mhealth-24-97. eCollection 2025. PMID 41211016

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT06985251/Prot_SAP_000.pdf